CLINICAL TRIAL: NCT01306903
Title: Minimal Extracorporeal Circuits (MECC) in Cardiac Surgery Procedures
Acronym: MECC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, Arndt-H. Kiessling, PI, Johann Wolfgang Goethe University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Mini-ECC001AHK
Record Dates: First submitted 2011-03-01; First posted 2011-03-02 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-06

CONDITIONS: Postoperative Bloodloss
Keywords: Minimizing Cardiopulmonary Bypass MECC damage organ failure
MeSH Terms: interventions — Chromatography, Micellar Electrokinetic Capillary

ARMS (3):
- MECC (Experimental): Minimal extracorporeal circuit
  Interventions: Device: MECC
- MOPS (Placebo Comparator)
  Interventions: Device: MOPS
- Super MOPS (Placebo Comparator)
  Interventions: Device: Super MOPS

INTERVENTIONS:
Device: MECC — Minimized extracorporeal circulation
  Arms: MECC
Device: MOPS — Modified and optimized perfusion system Frankfurt
  Arms: MOPS
Device: Super MOPS — Super modified and optimized perfusion system Frankfurt
  Arms: Super MOPS

SUMMARY:
The standard heart-lung machine is a major trigger of systemic inflammatory reactions, hemodilution, coagulopathy or organ failure. The strict reduction of blood-artificial surface and blood-air contact might represent meaningful improvements of the extracorporeal technology with respect to organ preservation.

The aim of this study is the evaluation of potential differences between a minimal extracorporeal circuit (MECC) and a conventional cardiopulmonary bypass (MOPS) system.

ELIGIBILITY:
Inclusion Criteria:

* extracorporeal circulation
* age > 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2011-03; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Bloodloss | postoperative
  Count of red blood packages

CONTACTS AND LOCATIONS:
Overall Officials: Arndt H Kiessling, MD, Principal Investigator — Goethe University Frankfurt
Locations (1):
- Goethe University Hospital, Frankfurt, Germany

REFERENCES:
- See also: Research THG — http://www.kgu.de/index.php?id=3615